CLINICAL TRIAL: NCT00700193
Title: An Open-Label, Multi-Centre Study to Evaluate the Safety, Tolerability and Immunogenicity of CSL's Influenza Vaccine in a Paediatric Population (= or >6 Months to < 9 Years of Age).
Brief Title: A Study of the Safety, Tolerability & Immunogenicity of CSL Limited's Influenza Virus Vaccine In a Paediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-FLU-04-05
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Equal to or greater 6 months to less than 3 years old
  Interventions: Biological: Influenza Virus Vaccine
- Group B (Other): Equal to or greater 3 years to less than 9 years old
  Interventions: Biological: Influenza Virus Vaccine

INTERVENTIONS:
Biological: Influenza Virus Vaccine — 2 dose vaccine regimen: 2 X 0.25mL vaccinations 30 days apart and a booster vaccination was administered 12 months after the first dose
  Arms: Group A
Biological: Influenza Virus Vaccine — 2 dose vaccine regimen: 2 X 0.50mL vaccinations 30 days apart and a booster vaccination was administered 12 months after the first dose
  Arms: Group B

SUMMARY:
The purpose of this study is to determine the Safety, Tolerability & Immunogenicity of CSL Limited's Influenza Virus Vaccine in a two dose primary vaccination series, with a 12-month booster vaccination, in a paediatric population equal to or greater than 6 months to less than 9 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Be healthy male or female children, aged = or > 6 months to < 9 years at the time of first study vaccination; Note: = or > 6 refers to 6 calendar months
2. Parent(s) or Guardian(s) to provide written informed consent to participate in the study;
3. Be able to provide a pre-vaccination sample of up to 5mL of venous blood without undue distress/discomfort and
4. Be born after a normal gestation period (between 36 and 42 weeks).

Exclusion Criteria:

1. Known allergy to eggs, chicken feathers, neomycin, polymyxin, or any components of the vaccine;
2. Previous influenza vaccination;
3. Clinical signs of active infection and/or an axillary temperature of = or >37.5 degrees Celsius or oral temperature of = or >38 degrees Celsius at study entry. Study entry may be deferred for such individuals, at the discretion of the Principal Investigator;
4. Confirmed or suspected immunosuppressive condition (including cancer), or a previously diagnosed (congenital or acquired) immunodeficiency disorder (including HIV);
5. Current (or within the 90 days prior to receiving the Study Vaccine) treatment with immunosuppressive or immunomodulative medication, including systemic corticosteroids, as follows:

   •Chronic or long term corticosteroids: >0.5mg/kg/day of oral prednisolone or equivalent (Note: Use of topical or inhalant corticosteroids prior to administration of the Study Vaccine or throughout the Study is acceptable).
6. Administration of immunoglobulins and/or any blood products since birth or planned administration of such blood products during the study period;
7. Participation in a clinical study or use of an investigational compound (ie a new chemical or biological entity not registered for clinical use), within the 90 days prior to receiving the Study Vaccine or be planning to enter such a study during the study period;
8. Current treatment with cytotoxic drugs or treatment within the 6 months prior to administration of the Study Vaccine;
9. Have a known history of Guillain-Barré Syndrome;
10. Have a major congenital defect or serious illness and
11. Have a history of neurologic disorders or seizures

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 298 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety of CSL Influenza Virus Vaccine in a Paediatric population through the assessment of the frequency of Local and general solicited symptoms, Unsolicited Adverse Events (UAE),Serious Adverse Events (SAEs) | Local & general solicited symptoms for 7 days post each vaccination, UAEs for 30 days post each vaccination, SAEs for 6 months after the last primary vaccination and 6 months after the booster vaccination

SECONDARY OUTCOMES:
Evaluate immunogenicity response to CSL Influenza Virus Vaccine in Paediatric population according to the criteria of the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines | 30 days after each vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Nolan, Prof, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Childrens Research Institute, Melbourne, Victoria, Australia